CLINICAL TRIAL: NCT03214523
Title: Freshman Sleep and Health Project
Acronym: FRoSH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17-0761
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Preventative Health; Sleep; Weight
Keywords: sleep; actigraphy
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Intervention Model Description: Half the subjects will be followed without any attempt to improve sleep, and half will undergo a brief educational intervention to try to improve sleep.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were recruited without emphasis on study arm. All outcomes will be assessed without knowledge of the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Education (Experimental): The intervention will be a brief education of the importance of sleep and healthy sleep habits. Subjects will also receive a standard sleep brochure on healthy sleep (which will also be given to the other arm).
  Interventions: Behavioral: Sleep Education
- Sleep Brochure (No Intervention): Subjects will receive a one page hand out on healthy sleep habits.

INTERVENTIONS:
Behavioral: Sleep Education — The subject will undergo a 30-minute session on sleep education from one of the study coordinators.
  Arms: Sleep Education

SUMMARY:
Sleep is a clearly necessary neurobiologic process that influences innumerable aspects of basic daily functions, physical health, and mental well-being. Recent literature shows that college students across the country are experiencing high rates of sleep deprivation. Interestingly, some recent studies have implicated this sleep loss in contributing to weight gain that occurs in the first year of college, also known as the "freshman fifteen." Rates of depression and other mental health issues, which are closely connected to sleep disturbances, are also on the rise in college campuses. The majority of the sleep data obtained in this population has been via questionnaires and self report, and the studies usually include college students at all seniority levels (e.g., freshmen, sophomores, seniors). Here, the investigators outline a novel study investigating how sleep time changes in college freshman, and how it relates to multiple different aspects of their health and functioning over the course of one quarter.

As technology has advanced, the ability to easily obtain objective measurements of different health parameters has increased dramatically. The investigators plan to use wireless actigraphy devices to measure sleep over a baseline seven day period in college-bound UCSD students prior to matriculation, and for 2 additional seven day periods during the first quarter of college. To the knowledge of the investigators, this is the first study to directly measure sleep time in college freshman in their normal environment. Effects of sleep time loss will be evaluated through multiple different metrics of physical and mental health. Given the recent link between sleep disturbances and weight gain in college freshman, the investigators will plan to measure weight changes prior to entering college and at two different time points through the first quarter. The investigators will use the PSQ-9 and GAD7 batteries as measures of mental health, obtained at the same time points as the sleep and weight information. As one of the primary consequences of sleep deprivation is on neurocognition in the daytime, the investigators plan to measure vigilant attention using psychomotor vigilance testing (PVT) as well. Screen time use has recently been targeted as a possible contributor to sleep loss in adolescents as well as adults and is something the investigators will attempt to measure as well using a smartphone application. Finally, this project will test the efficacy of a one hour sleep education intervention on improving total sleep time.

To the knowledge of the investigators, no other studies have closely examined how total sleep time changes during the first year of college in freshman in relationship to weight and mental health parameters, nor has PVT been done in this context. Additionally, with the increasing concerns regarding screen time use in adolescents and young adults, this study provides prime opportunity to examine this issue in the context of sleep.

ELIGIBILITY:
Inclusion Criteria:

* Incoming UCSD freshman

Exclusion Criteria:

* Under 18 years of age
* Not living on UCSD campus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Duration | Baseline, 4 weeks, 8 weeks
  Change in sleep duration pre and post-college start
Change in Weight | Baseline, 4 weeks, 8 weeks
  Change in weight pre and post-college start

SECONDARY OUTCOMES:
Symptoms of Depression | Baseline, 4 weeks, 8 weeks
  Symptoms of depression as assessed by standard questionnaire
Symptoms of Anxiety | Baseline, 4 weeks, 8 weeks
  Symptoms of anxiety as assessed by standard questionnaire
Reaction Time | Baseline, 4 weeks, 8 weeks
  Psychomotor vigilence testing

CONTACTS AND LOCATIONS:
Overall Officials: Robert Owens, MD, Principal Investigator — UCSD
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan at the current time to share data with other researchers.